CLINICAL TRIAL: NCT04209699
Title: An Open-label 3×3 Cross-over Study to Compare Effects of Famotidine Pretreatment and of Food on the Relative Bioavailability of Single Doses of BMS-986165 in Healthy Volunteers
Brief Title: A Study Comparing the Effects of Famotidine Pretreatment and of Food on the Relative Bioavailability of BMS-986165 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-119
Record Dates: First submitted 2019-12-23; First posted 2019-12-24 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib; Famotidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: BMS-986165 alone, fasted (Experimental)
  Interventions: Drug: BMS-986165
- Treatment B: BMS-986165 alone, fed (Experimental)
  Interventions: Drug: BMS-986165
- Treatment C: BMS-986165 with famotidine pretreatment, fasted (Experimental)
  Interventions: Drug: BMS-986165; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986165 — Single dose
Drug: Famotidine — Single dose
  Arms: Treatment C: BMS-986165 with famotidine pretreatment, fasted

SUMMARY:
The primary purpose of this study is to evaluate the effects of food and pH on the relative bioavailability (BA) of the tablet formulation of BMS-986165 in healthy volunteers

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body mass index of 18.0 kg/m^2 to 32.0 kg/m^2, inclusive, and body weight ≥ 50 kg, at screening
* Male and female paritcipants, aged 18 years, or age of majority, to age 55 years, inclusive
* All female subjects must have a negative serum or urine pregnancy test

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease.
* History of administration of live vaccines within 60 days before screening until clinic discharge
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population

Other protocol-defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for BMS-986165 for tablet dosed with high-fat high-calorie meal versus fasted condition | Day 1 to Day 13
Maximum observed plasma concentration (Cmax) for BMS-986165 for tablet administered fasted after pretreatment with famotidine vs administered alone | Day 1 to Day 13
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) in plasma for BMS-986165 for a tablet dosed with high-fat high-calorie meal versus fasted condition | Day 1 to Day 13
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) in plasma for BMS-986165 for tablet administered fasted after pretreatment with famotidine vs administered alone | Day 1 to Day 13
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) in plasma for BMS-986165 for tablet dosed with high-fat high-calorie meal versus fasted condition | Day 1 to Day 13
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) in plasma for BMS-986165 for tablet administered fasted after pretreatment with famotidine vs administered alone | Day 1 to Day 13

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 39 days
Number of clinically significant changes in vital sign measurements | Up to 18 days
Number of clinically significant changes in clinical laboratory test results | Up to 18 days
Number of clinically significant changes in electrocardiogram (ECG) parameters | Up to 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm